CLINICAL TRIAL: NCT01392248
Title: EEG as a Predictor for Postoperative Pain and the Development of Chronic Postsurgical Pain After Breast Cancer Surgery
Brief Title: Prediction of Pain After Breast Cancer Surgery With EEG
Status: Terminated | Type: Observational
Why Stopped: funding and recruiting problems
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Carine Vossen, MD, Maastricht University Medical Center
Other Study IDs: NL34275.068.11 / MEC 11-2-006
Record Dates: First submitted 2011-06-01; First posted 2011-07-12 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Breast Cancer; Postoperative Pain; Chronic Pain
Keywords: EEG; breast cancer surgery; prediction; acute postoperative pain; chronic pain
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
1. Rationale The inter-individual pain experience immediately after surgery is considerable. In addition, a number of patients develop chronic post surgery pain (CPSP). Patients undergoing surgery for breast cancer are at risk of developing both acute post surgical pain as well as CPSP. Recently, in a group of patients with chronic back pain, it was demonstrated how subjectively reported pain is associated with specific electroencephalography (EEG) parameters, namely the N2 and P3 components of the pain event-related potential (ERP). It was concluded that ERP was associated with self-reported pain in daily life up to two weeks after the measurement. This resulted in the current hypothesis that EEG may be a predictor for postoperative pain.
2. Study design Prospective cohort study. Within 2 weeks before surgery, 150 patients will undergo an EEG measurement with five 'vulnerability' tasks. The experiment will be repeated 6 months postoperatively.

   Study population: Female patients with breast cancer who will undergo breast surgery, between the ages of 18 to 65 years.
3. Main study parameters/endpoints Primary outcome is postoperative pain, measured in a pain diary 4 days postoperatively. Secondary outcomes are development of chronic post surgery pain and quality of life. The main goal is to develop a comprehensive prediction model for acute and chronic postoperative pain after breast cancer surgery, based on the EEG results of the five vulnerability experiments.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 65 years.
* ASA 1-2.
* Sufficient comprehension of the Dutch spoken and written language.
* Elective curative breast cancer surgery, both mastectomy and breast- conserving therapy
* Stage I and II breast cancer.
* Written informed consent is obtained

Exclusion Criteria:

* Previous breast surgery, both ipsilateral and contralateral.
* Stage III-IV breast cancer.
* Chronic pain (>3months) with an average severity of at least a VAS score 4 during the last two weeks.
* Chronic pain for which invasive treatment is needed.
* Use of (weak / strong) opioids in the last week.
* A history of opioid addiction.
* Regular use of the following medications in the last year:

antiepileptics,antipsychotics and anxiolytics.

* ASA 3 or higher.
* Consumption of alcohol (>4 units) and / or drugs the evening before.
* Alcohol consumption (>= 5 units/day).
* Illiteracy, problems with self expression, language barrier.
* Serious vision and / or hearing problems, interfering the performance of the experimental tasks.
* A history of psychiatric complaints and/or epilepsy .
* A medical history of CVA or TIA.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One hundred and fifty female patients undergoing elective breast cancer surgery in day-case surgery.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2011-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Acute postoperative pain | during 4 days after surgery
  VAS measured in a daily pain diary

SECONDARY OUTCOMES:
Quality of Life | within 2 weeks before surgery and at 3,6 and 12 months postoperatively
  Quality of Life measured with SF-36
Development of chronic pain | at 3,6 and 12 months postoperatively
  Brief Pain Inventory

CONTACTS AND LOCATIONS:
Overall Officials: M. A Marcus, Prof. Dr., Principal Investigator — Maastricht University Medical Center; J. van Os, Prof. Dr., Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht UMC, Maastricht, Limburg, Netherlands